CLINICAL TRIAL: NCT02918123
Title: Phase 1 Clinical Trial to Evaluate the Safety of FURESTEM-CD Inj. in Patients With Moderate to Severe Plaque-type Psoriasis.
Brief Title: Safety of FURESTEM-CD Inj. in Patients With Moderate to Severe Plaque-type Psoriasis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kang Stem Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSB-PsO
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Psoriasis
Keywords: Psoriasis; Plaque psoriasis; Stem cell; Cell therapy; Furestem; Mesenchymal stem cell; MSC; Umbilical cord blood; hUCB-MSC; UCB-MSC
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): 1. FURESTEM-CD Inj. 5.0x10^7 cells
  2. FURESTEM-CD Inj. 1.0x10^7 cells
  3. FURESTEM-CD Inj. 2.0x10^8 cells
  Interventions: Biological: FURESTEM-CD Inj.

INTERVENTIONS:
Biological: FURESTEM-CD Inj. — Patients will be treated FURESTEM-CD Inj. Subcutaneous injection
  Other Names: hUCB-MSCs

SUMMARY:
Phase I clinical trial to evaluate safety of FURESTEM-CD Inj. in patients with moderate to severe in plaque-type psoriasis injection for 4weeks.

DETAILED DESCRIPTION:
This is a phase 1, single center, randomized, open label, study of safety of FURESTEM-CD Inj. in subjects with moderate to severe plaque psoriasis.

Approximately 9~18 subjects will be administrated FURESTEM-CD Inj.

FURESTEM-CD Inj. is composed of allogeneic hUCB-MSC(human Umbilical Cord Blood derived-Mesenchymal Stem cell). hUCB-MSCs are mesenchymal stem cells from umbilical cord blood. Mesenchymal stem cells are well-known for immunosuppression, anti-inflammatory ability and capable of differentiating into a wide range of cell types. Therefore, FURSTEM-CD Inj. has huge possibility as cell therapy products for plaque-type Psoriasis patients.

ELIGIBILITY:
Inclusion Criteria:

1. 19-65 years old(both sexes)
2. Have been diagnosed with plaque-type psoriasis at least 6 months prior to screening (subjects with concurrent psoriatic arthritis[PsA] may be enrolled)
3. Psoriasis Area and Severity Index (PASI) score >= 12 at screening
4. BSA(Body Surface Area) >= 10 percentage at screening
5. Have had at least one of the following conventional systemic agent for the treatment of psoriasis,

   * MTX, Cyclosporine, Photochemotherapy, TNF-alpha inhibitor or IL-12/IL-23 inhibitor
6. Subject who would agree to avoid prolonged sun exposure, use of tanning booths or other ultraviolet light sources during the clinical study
7. Subject who understands and voluntarily signs the informed consent form

Exclusion Criteria:

1. Subject who has other types of psoriasis (eg. Erythrodermic, guttate, or pustular)
2. Have a history of chronic or recurrent infectious disease
3. Have received phototherapy or any systemic medications/treatments within 4 weeks of screening that could affect psoriasis or PASI evaluation
4. Have used topical medications/treatments within 2 weeks of screening that could affect psoriasis or PASI evaluation
5. Have used any systemic immunosuppressants within 4 weeks of screening
6. Have been administered with the following biological agents that could affect plaque-type psoriasis

   * Etanercept - within 4 weeks of screening
   * Adalimumab, alefacept, infliximab - within 2 months of screening
   * Ustekinumab - within 4 weeks of screening
   * Other investigational biological agents - within 4 weeks of screening/five half-lives(whichever was longer)
7. Pregnant, breast-feeding women or women who plan to become pregnant during this study (Females of childbearing potential must have a negative urine pregnancy test at screening)
8. Have been administered any types of investigational drugs within the previous 4 weeks or five half-lives of the investigational agent, whichever is longer
9. Subject who already took or need to take medicine which is prohibited during the clinical study
10. Subject who has sever dyshepatia (Creatinine value ≥ 2X Upper limit of the normal range at screening test)
11. Subject who has severe renal dysfunction (AST/ALT value ≥ 2X Upper limit of the normal range at screening test)
12. Have received a live viral or bacterial vaccination within 3 months of screening
13. Have had a BCG(Bacillus Calmette-Guérin) vaccination within 12 months of screening
14. Have a transplanted organ(with the exception of a corneal transplant > 3 months prior to screening)
15. Have any known malignancy or have a history of malignancy
16. Have a history of hypersensitivity, heavy metal poisoning etc. to drugs which are composed of similar components or have undergone allergy immunotherapy previously for prevention of anaphylactic reactions
17. Have had a serious infection (eg. Sepsis, pneumonia or pyelonephritis), or have been hospitalized or received IV antibiotics for an infection during the 2 months prior to screening
18. Positive for Hepatitis B virus(HBV) surface antigen or anti-Hepatitis C virus antibody screening
19. Known to have had a substance abuse(drug or alcohol) problem within 12 months of screening
20. Subject who experienced stem cell therapy
21. Any other conditions which the PI suspect the patient to be unsuitable for the clinical

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2018-01-17 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
number of adverse events | 4 weeks follow-up after treatment
safety lab tests, physical examination, ECG, vital signs | 4 weeks follow-up after treatment
variation of Cytokine, PASI, BSA | 4 weeks follow-up after treatment

OTHER OUTCOMES:
number of adverse events, safety lab tests, physical examination, vital signs | 144 weeks follow-up after treatment (Extension study)

CONTACTS AND LOCATIONS:
Overall Officials: Taeyoon Kim, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- The Catholic Univ. Korea Seoul, St. Marry's Hospital, Seoul, South Korea